Title of the study:

# Influence of human platelet derivatives on dental implant.

Study Number:

**MUOSU-202103.** 

Date: 7/9/ 2023

day / month / year



# RESEARCH ETHICS: PATIENT INFORMATION FORM

Study Number: MUOSU-202103

Title of Project: Influence of human platelet derivatives on dental implant.

# Principle investigator: Dr. Afya Sahib Diab

# 1- What is the purpose of this study?

To develop the science of dental Implantology and find new ways to increase the success rates of dental implants

#### 2- Why have I been chosen?

You have missing teeth and you need dental implants to replace the missing teeth.

#### 3- Do I have to take part?

No, it's up to you

#### 4- What will happen to me if I take part?

Nothing will happen to you except you are going to help me carrying out my study research

#### 5- What are the possible disadvantages and risks of taking part?

There is no possible risk or disadvantage of taking part

## 6- What are the possible benefits of taking part?

Taking part will facilitate my work during the research by collecting required number of cases needed which may provide beneficial treatment alternatives for you as well as others in the future

### 7- Will my taking part in this study be kept confidential?

Sure, your information will be kept private

#### 8- What will happen to the results of the research study?

The results of the study research will be published in scientific magazines for the benefit of all

#### 9- Who is organizing & hosting the research?

Mustansiriyah University / College of dentistry

#### 10- What if I need more information about the way in which this study has been conducted?

You can ask your dentist about any information you need

Principal investigator: Dr. Afya Sahib Diab

Email: drafya\_diab@yahoo.com Phone No. +964(0)7816883387

| Study Number: MUOSU-202103 | | we die die de la company de la |
|---|---|---|
| Patient identification number for t | his study: | 3000 |
| | | Louis Comit |
| | Consent form | |
| Title of the Project: Influence of human platelet derivatives on dental implant | | |
| Principle investigator: Dr. Afya S | Sahib Diab | |
| 2. I understand that my participation is vol | luntary and that I am free to | withdraw at any time |
| I confirm that I have read and understated opportunity to consider the information. | | · |
| without giving any reason, without my | y medical care or legal rights | s being affected. |
| 3. I understand that relevant sections of r may be looked at by individuals from repart in this research. I give permission | egulatory authorities, where | it is relevant to my taking |
| . further samples may be taken during dent<br>time stage of treatment. | tal treatment as patients are l | being recruited at different |
| I agree to take part in the above s | study | |
| Name of the participant | Date: day / month/ year | Signature |
| Name of person taking consent | Date: day / month/ year | Signature |